CLINICAL TRIAL: NCT00071188
Title: A Randomized, Partially Blinded, Phase II Study to Assess the Safety, Tolerability and Efficacy of ZD6474 Alone or in Combination With Paclitaxel and Carboplatin in Subjects With Previously Untreated Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: ZD6474 Alone or in Combination With Paclitaxel and Carboplatin in Subjects With Previously Untreated Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00007; D4200C00007(run-in); D4200C0007A (randomization); NCT00093392 (obsolete NCT alias)
Record Dates: First submitted 2003-10-14; First posted 2003-10-16 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: ZD6474
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The purpose of the run-in phase of this study is to determine the appropriate and tolerable dose of ZD6474 (200mg or 300mg) to be administered in combination with paclitaxel and carboplatin in subjects with previously untreated locally advanced or metastatic NSCLC. This phase of the trial is closed to enrollment.

The purpose of the randomized phase of this study is to determine the efficacy of ZD6474 alone versus that of ZD6474 in combination with paclitaxel and carboplatin versus that of paclitaxel and carboplatin alone in subjects with previously untreated locally advanced or metastatic NSCLC. This phase of the trial is closed to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years or older
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC
* No prior chemotherapy/biological therapy/radiation therapy
* One or more measurable lesions
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Brain metastases or spinal cord compression
* Currently active skin disease
* History of significant hemoptysis
* Abnormal blood chemistry
* Cardiac abnormalities
* Recent significant cardiac event
* Coexisting malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (34):
- United States (12):
  - Research Site, Concord, California
  - Research Site, Los Angeles, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Turku
- France (3):
  - Research Site, Besançon
  - Research Site, Lille
  - Research Site, Strasbourg
- Germany (4):
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Mainz
  - Research Site, Ulm
- Research Site, Pune, India
- Italy (2):
  - Research Site, Milan
  - Research Site, Orbassano
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Panorama
  - Research Site, Parkland
  - Research Site, Pretoria
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
- Research Site, Chiang Mai, Thailand